CLINICAL TRIAL: NCT05497752
Title: Effectiveness of Cervical Rehabilitation Program on Neck Pain, ROM and Disability After Thyroidectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Tayyaba Sultan
Record Dates: First submitted 2022-08-10; First posted 2022-08-11 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Thyroiditis, Postpartum
Keywords: positional release; suboccipital muscle release
MeSH Terms: conditions — Postpartum Thyroiditis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical rehabilitation group (Experimental): Positional release technique on trapezius muscle, suboccipital muscle release, pectoralis muscle stretching
  Interventions: Other: cervical rehabilitation program
- control group (Active Comparator): shoulder and neck exercises
  Interventions: Other: control group

INTERVENTIONS:
Other: cervical rehabilitation program — (Positional release technique on trapezius muscle): The subject was supine The therapist applied Pressure by pinching the trapezius muscle between the thumb and fingers.
  Suboccipital muscle release):
  The patient will be in a Supine lying position therapist places both his palms at suboccipital region with upward pressure causing a stretch and distraction for 30 seconds. This technique was performed 3 times in one session with a rest interval of 1 minute after each time.
  (Stretching of pectoralis muscle):. once daily Stretching with repetition of five, three times a day for 1week
  Arms: cervical rehabilitation group
Other: control group — Relax shoulders and neck sufficiently look down turn face to the right turn face to the left incline head to the right incline head to the left turn shoulders round and round slowly raise hands fully then lower them. patients were asked to perform five repetitions of each stretching exercise, three times per day (morning, afternoon, and evening).
  Arms: control group

SUMMARY:
The aim of this research is to determine the Effects of cervical rehabilitation program on neck pain, ROM and disability after thyroidectomy. Randomized controlled trials will be done at Pakistan ordinance factory (POF) Hospital. The sample size will be 52. The subjects were divided in two groups, with 26 subjects in Group A and 26 in Group B. Study duration will be of 6 months. Sampling technique applied will be Non probability Convenience Sampling technique. Both males and females of aged 30-50 years with thyroidectomy will be included. Tools used in the study are Numeric Pain Rating Score (NPRS), goniometer and neck disability index (NDI).

DETAILED DESCRIPTION:
Thyroidectomy, or surgical removal of the gland, is highly recommended treatment for thyroid disorders. The most prevalent of these conditions are symptomatic benign large goiter and tumorous condition of the thyroid gland. Both younger females and postmenopausal older women are prevalent towards these disorders (nodular goiter, cancer, and hypothyroidism).

Due to hyperextended position of neck during surgery patient usually complaint about the posterior neck pain, movement difficulties of shoulder and neck, occipital headaches, shoulder stiffness, motion's cervical range of limitations and some of them experiences the discomfort symptoms such as stretching, pressing, or choking feelings in the neck, headache, shoulder stiffness, and difficulty in moving the neck or shoulders. These symptoms may persist for an extended period following surgery and may even have a negative effect on the patient's quality of life. It has been reported that hyperextension can cause bilateral hypoglossal palsy, tetraplegia and cervical artery dissection.

Recently, a variety of treatment modalities have been used to overcome these disturbing symptoms, such as intraoperative transcutaneous electrical nerve stimulation (TENS), preoperative bilateral greater occipital nerve (GON) block, bilateral superficial cervical plexus block combined with bilateral GON block, and postoperative neck stretching exercise. Due to surgical position of thyroidectomy patient often develops posture syndrome of thyroid surgery (PSTS), symptoms include postoperative nausea, vomiting, dizziness, headache and some discomfort associated with neck an occipital radiating pain.

Position of neck during surgery and static posture of patient after thyroidectomy causes tightness of surrounding muscles which leads to posterior neck pain, limited ROM and functional disability. Everyone is focused on the incisional pain but not on this disability, there is some literature on neck stretching exercises to treat posterior neck pain but no other technique is used for treatment of posterior neck pain. The purpose of this study is to check the effectiveness of cervical rehabilitation program on neck pain, ROM and disability following thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* • Both genders (male & female)

  * Post-thyroidectomy patients
  * Indoor patients

Exclusion Criteria:

* • Any cervical fracture/dislocations

  * Cervical instability
  * Vertebrobasilar insufficiency
  * Cervical Radiculopathy
  * Disc prolapsed at cervical region
  * Any neurological impairment

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
NPRS | 1 Week
  It used to assess neck pain intensity. Patients were asked to rate how bad their neck pain will on average (NPRS; range, 0, no pain, to 10, maximum pain). pain will be assessed at baseline and after 1 week.
Neck disability index | 1 week
  is used to asses that how neck pain affects the quality of life of a person. It consists of 10 items, from 0-5 points in each item. Total score of NDI is 50 that is converted into percentage of 100 latterly.
  0-4 points (0-8%) no disability, 5-14 points ( 10 - 28%) mild disability, 15-24 points (30-48% ) moderate disability, 25-34 points (50- 64%) severe disability, 35-50 points (70-100%) complete disability

SECONDARY OUTCOMES:
neck flexion ROM | 1 week
  Goniometer is a tool used to assess the range of motion. The range of motion from neutral position to forward movement will be measured. reading will be taken at baseline and at 1st week.
neck Extension ROM | 1 week
  Goniometer is a tool used to assess the range of motion. The range of motion from neutral position to backward movement will be measured. reading will be taken at baseline and at 1st week.
neck Rt side flexion ROM | 1 week
  Goniometer is a tool used to assess the range of motion. The range of motion from neutral position to Rt side, ear towards the shoulder movement will be measured. reading will be taken at baseline and at 1st week.
neck Lt side flexion ROM | 1 week
  Goniometer is a tool used to assess the range of motion. The range of motion from neutral position to Lt side, ear towards the shoulder movement will be measured. reading will be taken at baseline and at 1st week.
neck Rt Rotation ROM | 1 week
  Goniometer is a tool used to assess the range of motion. The range of motion from neutral position to Rt side, Face towards the Rt side movement will be measured. reading will be taken at baseline and at 1st week.
neck Lt Rotation ROM | 1 week
  Goniometer is a tool used to assess the range of motion. The range of motion from neutral position to Rt side, face towards the Lt side movement will be measured. reading will be taken at baseline and at 1st week.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Heavy Industrial Taxila Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No